CLINICAL TRIAL: NCT03594266
Title: Comparison of the Effects of Two Spinal Cord Stimulation (SCS) Therapies on Subject Reported Pain (BENEFIT-02)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BENEFIT-02
Record Dates: First submitted 2018-07-09; First posted 2018-07-20 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Chronic Low Back Pain; Chronic Leg Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Therapy A Spinal Cord Stimulation Parameter Set (Experimental)
  Interventions: Device: Therapy A spinal cord stimulation parameter set using BIO-RNA system and associated components
- Therapy B Spinal Cord Stimulation Parameter Set (Experimental)
  Interventions: Device: Therapy B spinal cord stimulation parameter set using BIO-RNA system and associated components

INTERVENTIONS:
Device: Therapy A spinal cord stimulation parameter set using BIO-RNA system and associated components — Therapy A stimulation patterns
  Arms: Therapy A Spinal Cord Stimulation Parameter Set
Device: Therapy B spinal cord stimulation parameter set using BIO-RNA system and associated components — Therapy B stimulation patterns
  Arms: Therapy B Spinal Cord Stimulation Parameter Set

SUMMARY:
A BIOTRONIK wearable stimulator will be utilized in order to investigate the effects of two study spinal cord stimulation (SCS) therapies on subject reported pain and paresthesia perception observed over 12 days of study stimulation testing following the conclusion of a successful SCS commercial trial.

DETAILED DESCRIPTION:
The study population will consist of patients with chronic low back and/or leg pain who have been identified as candidates for trial testing of a commercially available SCS system including percutaneous SCS trial lead(s), but have not yet undergone trial lead implant. The commercial trial test period will be conducted independently from the study according to standard of care. The commercial trial period is referred to as the "trial" and the BENEFIT-02 interventional study stimulation period is referred to as the "study".

Potential subjects will be identified by the investigator from their general patient population and must meet all of the study inclusion and none of the study exclusion criteria evaluated at the time of enrollment. Once study eligibility is confirmed, written informed consent is obtained, after which enrollment visit data will be collected. Subjects will be considered fully enrolled after being randomly assigned to receive one of two study SCS therapies.

To participate in this study, subjects must be willing to undergo an extended 14 day testing period following the conclusion of their commercial trial, where their existing SCS trial lead(s) will be connected to a BIOTRONIK study stimulator and one of two randomly assigned study SCS therapies will be administered for an additional 12 days after a two day washout period. After completion of the 12 day study testing period, the subject's participation in the study ends, the study stimulator will be disconnected, and the commercial SCS trial lead(s) will be removed according to the standard clinical routine.

This feasibility study includes the assessment of two primary endpoints and two secondary endpoints that are designed to provide preliminary information regarding the effectiveness and safety of the two study SCS therapies under investigation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Able to understand the nature of the study and provide written informed consent
* Able to read, understand, and speak English
* Willing and able to comply with all study requirements, including all required procedures, phone calls and study visits
* Planned to undergo a commercial SCS trial of standard duration for the treatment of low back and/or leg pain with a commercially available SCS system as prescribed by a physician(s) according to FDA approved indications for use
* Planned utilization of preoperative antibiotics for SCS commercial trial
* Planned placement of two eight-electrode SCS trial leads (or at least one 16- electrode SCS trial lead) using a suitable technique for an extended trial (e.g. tunneling approach of a minimum of 3-4 cm, or buried lead trial) with at least one lead covering the T8 or T9 vertebral level
* Incoming Numerical Rating Scale (NRS) for pain (overall) of at least 6 (collected prior to the commercial trial)
* Passed psychological evaluation
* Negative MRSA screening result
* Negative MSSA screening result or documentation of subsequent decolonization routine if MSSA positive
* For diabetic patients: minimum of one HbA1c test within the last 6 months, with most recent result ≤ 7.5%

Exclusion Criteria:

* Enrolled in any investigational SCS stimulation trial, for which the SCS system is not commercially available
* Presence of any life-threatening, underlying illness separate from their indication for SCS therapy
* Patients reporting pregnancy at the time of enrollment
* Patients with poor compliance for pain management regimen
* Patients currently involved in an active workers compensation claim and/or active litigation related to injury associated with indication for SCS
* Patients with a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency (other than prescribed) in the 6 months prior to baseline data collection
* Patients with an implanted pacemaker, defibrillator, or other medical contraindications for SCS therapy
* Patients with a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the investigator
* Patients immunocompromised and/or at high risk for infection
* Patients with morphine equivalent dose > 120 units
* Patients with documented history of allergic response or sensitivity to material(s) required for the study (e.g. silver impregnated antibacterial dressing, adhesives, titanium, silicone, etc.)
* Patients with a documented history of clostridium difficile

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Kapural, MD, Study Chair — Carolinas Pain Institute
Locations (18):
- United States (18):
  - Hope Research Institute, Peoria, Arizona
  - Arizona Pain, Scottsdale, Arizona
  - Integrated Pain Management (IPM) Medical Group, Walnut Creek, California
  - Center for Interventional Pain and Spine, Wilmington, Delaware
  - Coastal Orthopedics, Bradenton, Florida
  - Pain Care, LLC, Stockbridge, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - Neuroscience Research Center DBA Kansas Pain Management, Overland Park, Kansas
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - St. Louis Pain Consultants, Chesterfield, Missouri
  - KC Pain Centers, Lee's Summit, Missouri
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Ainsworth Institute of Pain Management, New York, New York
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Integrated Pain Solutions, Columbus, Ohio
  - Delaware Valley Pain and Spine Institute, Trevose, Pennsylvania
  - Northwest Pain Care, Inc., Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapural L, Patterson DG, Li S, Hatheway J, Hunter C, Rosen S, Fishman M, Gupta M, Sayed D, Christopher A, Burgher A, McJunkin T, Ross EL, Provenzano D, Amirdelfan K. Multiphase Spinal Cord Stimulation in Participants With Chronic Back or Leg Pain: Results of the BENEFIT-02 Randomized Clinical Trial. Neuromodulation. 2023 Oct;26(7):1400-1411. doi: 10.1016/j.neurom.2023.05.006. Epub 2023 Aug 16. PMID 37589641

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 136 provisionally enrolled participants, 77 met the criteria to be randomized to treatment.
Groups:
- Therapy A Spinal Cord Stimulation Parameter Set: Therapy A (~600-1500Hz) spinal cord stimulation parameter set using BIO-RNA system and associated components.
- Therapy B Spinal Cord Stimulation Parameter Set: Therapy B (~300-600Hz) spinal cord stimulation parameter set using BIO-RNA system and associated components.
Period: Overall Study
Arm/Group | Therapy A Spinal Cord Stimulation Parameter Set | Therapy B Spinal Cord Stimulation Parameter Set
Started | 38 | 39
Completed | 31 | 34
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Enrolled But Not Randomized: Subjects selected for participation from the investigator's patient population who have signed the Informed Consent Form, have confirmation of the initial enrollment criteria, and have completed baseline measurements, but did not meet criteria to be randomized at office visit 1.
- Therapy A: Subjects meeting all eligibility criteria at office visit 1 and are subsequently randomized to Therapy A (~600-1500Hz) spinal cord stimulation parameter set.
- Therapy B: Subjects meeting all eligibility criteria at office visit 1 and are subsequently randomized to Therapy B (~300-600Hz) spinal cord stimulation parameter set.
- Total: Total of all reporting groups
Arm/Group | Enrolled But Not Randomized | Therapy A | Therapy B | Total
Number analyzed (Participants) | 59 | 38 | 39 | 136
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (12.09) | 60.8 (13.25) | 60.4 (13.79) | 62 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 24 | 82
  Male | 26 | 13 | 15 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 5
  Not Hispanic or Latino | 49 | 32 | 33 | 114
  Unknown or Not Reported | 7 | 5 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 4 | 15
  White | 45 | 31 | 33 | 109
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 1 | 9
Clinical Characteristics - Primary Pain Diagnosis [Count of Participants; unit: Participants] — Subject medical history characteristics collected for the study at time of enrollment.
  Participants
    Failed back surgery syndrome | 16 | 13 | 11 | 40
    Radiculopathy | 9 | 8 | 7 | 24
    Complex regional pain syndrome | 8 | 4 | 4 | 16
    Chronic pain syndrome | 5 | 3 | 6 | 14
    Degenerative disc disease | 5 | 3 | 3 | 11
    Spinal stenosis | 4 | 2 | 3 | 9
    Low back pain | 3 | 1 | 4 | 8
    Dorsalgia | 2 | 1 | 1 | 4
    Spondylosis | 2 | 0 | 0 | 2
    Other primary pain diagnosis | 3 | 2 | 0 | 5
    Unknown primary pain diagnosis | 2 | 1 | 0 | 3
Clinical Characteristics - Previous Back Surgery [Count of Participants; unit: Participants]
  Yes | 31 | 25 | 25 | 81
  No | 27 | 13 | 14 | 54
  Unknown | 1 | 0 | 0 | 1
Clinical Characteristics - Taking Opioid Analgesics [Count of Participants; unit: Participants]
  Yes | 34 | 19 | 21 | 74
  No | 22 | 19 | 18 | 59
  Unknown | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change Since Baseline in Numerical Rating Scale (NRS) for Pain (Overall) Evaluated Separately for Each Study SCS Therapy
Description: The purpose of primary endpoint 1 is to evaluate the change since baseline in Numerical Rating Scale (NRS) for pain (overall) for each study SCS therapy. The evaluation of primary endpoint 1 is based on the NRS for pain (overall) obtained at the final study testing visit compared with the baseline measurement obtained prior to initiation of the commercial trial period, for subjects randomized to each study SCS therapy. Numerical Rating Scale (NRS) was collected for overall pain experienced over the past 24 hours on a scale of 0-10, with 0 being No Pain and 10 being Worst Possible Pain.
Time Frame: Baseline and in-office visit 3, average of 21 days
Population: Only patients with valid NRS for pain (overall) at both baseline and at in-office visit 3 were evaluated for this endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Therapy A Spinal Cord Stimulation Parameter Set | Therapy B Spinal Cord Stimulation Parameter Set
Number analyzed (Participants) | 24 | 23
Score on a scale | -4.3 (0.47) | -4.7 (0.48)
Statistical Analysis 1: Comparison: Therapy A Spinal Cord Stimulation Parameter Set; Test type: Other; p < 0.0001, paired t-test, two-sided
Statistical Analysis 2: Comparison: Therapy B Spinal Cord Stimulation Parameter Set; Test type: Other; p < 0.0001, paired t-test, two-sided

2. Primary Outcome: Inter-therapy Comparison of Change Since Baseline in Numerical Rating Scale (NRS) for Pain (Overall)
Description: The purpose of primary endpoint 2 is to provide an inter-therapy comparison of change since baseline in Numerical Rating Scale (NRS) for pain (overall). Primary endpoint 2 analyses includes all participants included in primary endpoint 1 analyses. Numerical Rating Scale (NRS) was collected for overall pain experienced over the past 24 hours on a scale of 0-10, with 0 being No Pain and 10 being Worst Possible Pain.
Time Frame: Baseline and in-office visit 3, average of 21 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Therapy A Spinal Cord Stimulation Parameter Set | Therapy B Spinal Cord Stimulation Parameter Set
Number analyzed (Participants) | 24 | 23
Score on a scale | -4.3 (0.47) | -4.7 (0.48)
Statistical Analysis 1: Comparison: Therapy A Spinal Cord Stimulation Parameter Set vs Therapy B Spinal Cord Stimulation Parameter Set; Test type: Other; p = 0.5482, two-sample t-test, 2-sided

3. Secondary Outcome: Change Since Conclusion of Commercial Trial in Numerical Rating Scale (NRS) for Pain (Overall) Evaluated Separately for Each Study SCS Therapy
Description: The evaluation of secondary endpoint 1 will be based on Numerical Rating Scale (NRS) for overall pain experienced over the past 24 hours (scale of 0-10, with 0 being No Pain and 10 being Worst Possible Pain) obtained at conclusion of commercial trial compared to NRS for overall pain at the final study testing visit
Time Frame: In-office visit 1 at approximately 7 days and in-office visit 3 at approximately 21 days, average of 14 days
Population: Only patients with valid NRS for pain (overall) at both in-office visit 1 and in-office visit 3 were evaluated for this endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Therapy A Spinal Cord Stimulation Parameter Set | Therapy B Spinal Cord Stimulation Parameter Set
Number analyzed (Participants) | 24 | 23
Score on a scale | 1.0 (0.53) | 0.3 (0.32)

4. Secondary Outcome: Investigational Device-related Adverse Event-free Rate
Description: The evaluation of secondary endpoint 2 will be based on the number of subjects free from investigational device-related adverse events assessed at in-office visit 1 (randomization visit) through in-office visit 3 (study completion). The investigational device-related adverse event-free rate was pre-defined within the protocol as the overall rate from all implanted Prospera SCS devices, regardless of randomized therapy output setting (Therapy A or Therapy B).
Time Frame: Baseline and in-office visit 3, average of 21 days
Population: Evaluable subjects for secondary endpoint 2 will include all subjects who undergo randomization and have the investigational stimulation system connected to their SCS trial leads. The investigational device-related adverse event-free rate was pre-defined within the protocol as the overall rate from all implanted Prospera SCS devices, regardless of randomized therapy output setting (Therapy A or Therapy B). Therefore, data for Therapy A and Therapy B are combined for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Provisionally Enrolled: Subjects were selected for participation from the investigator's patient population and are considered provisionally enrolled upon signing the Informed Consent Form and confirmation of the initial enrollment criteria. Provisionally enrolled subjects who meet all clinical eligibility criteria and have been randomized are considered fully enrolled.
Arm/Group | Subjects Provisionally Enrolled
Number analyzed (Participants) | 77
Participants | 76

ADVERSE EVENTS:
Time Frame: 21 days
Groups:
- Enrolled But Not Randomized: Subjects selected for participation from the investigator's patient population who have signed the Informed Consent Form and have confirmation of the initial enrollment criteria but have not yet been randomized.
- Therapy A: Subjects meeting all eligibility criteria who have been randomized to the Therapy A (~600-1500Hz) spinal cord stimulation parameter set.
- Therapy B: Subjects meeting all eligibility criteria who have been randomized to the Therapy B (~300-600Hz) spinal cord stimulation parameter set.
Arm/Group | Enrolled But Not Randomized | Therapy A | Therapy B
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 2/59 | 3/38 | 3/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled But Not Randomized (N=59) | Therapy A (N=38) | Therapy B (N=39)
Irritation from wound dressing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — SCS Trial Lead Implant Procedure-Related
Lead migration (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — SCS Trial Lead Implant Procedure-Related
Reaction from wound dressing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — SCS Trial Lead Implant Procedure-Related
Persistent post-surgical site pain (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Commercial Trial Period Related
Reaction from wound dressing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — Commercial Trial Period Related
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Commercial Trial Period Related
Neurostimulator device entered "safe mode" (Product Issues) | 0 (0) | 1 (1) | 0 (0) — Unknown Relationship to the Investigational Device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03594266/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT03594266/SAP_001.pdf